CLINICAL TRIAL: NCT05911958
Title: Phase II Study of SHR-A1811 as Neoadjuvant Treatment for Patients With HR-Positive, Low HER2 Expression Breast Cancer
Brief Title: A Study of SHR-A1811 as Neoadjuvant Treatment for Patients With HR-Positive, Low HER2 Expression Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Zhenzhen Liu, Professor, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HELEN-015; BC-NEO-IIT-SHR-A1811 (Other: Jiangsu Hengrui Medicine Co.,Ltd.)
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: HER2 Low Breast Carcinoma
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-A1811 (Experimental): SHR-A1811 group
  Interventions: Drug: SHR-A1811 for injection

INTERVENTIONS:
Drug: SHR-A1811 for injection — SHR-A1811 for injection
  Other Names: SHR-A1811 group

SUMMARY:
HR-positive breast cancers accounts for about 50% to 60% of all breast cancer patients. Neoadjuvant Chemotherapy is the core treatment mode for this type of breast cancer, and endocrine therapy can be used in some low-risk patients. However, the pathological complete response (pCR) rate obtained is low. HER2 is an important prognostic indicator and therapeutic target for breast cancer. Nearly 60% of HR-positive breast cancers have low expression of HER2, and antibody-drug conjugates (ADC) targeting HER2 may achieve better efficacy in this subtype.

DETAILED DESCRIPTION:
This prospective, single-arm study is being conducted to evaluate the efficacy and safety of SHR-A1811 for early-stage or locally advanced breast cancer patients with HR-Positive, Low HER2 Expression. Subjects will receive the neoadjuvant therapy of SHR-A1811 for eight cycles, and then undergo surgery within 4 weeks after neoadjuvant therapy. The follow-up visit will last for at least 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 70 years old (inclusive);
2. Treatment-naive patients with clinically confirmed T2-T3, any nodal status and M0;
3. HR-positive, HER2 low expression, the expression of Ki-67 exceed 14% invasive breast cancer confirmed by histology or cytology;
4. ECOG performance status of 0-1;
5. Normal organ and bone marrow function;
6. Patients of childbearing age must consent to use highly effective contraception for 7 months from the start of study screening until the last study medication and agree not to breastfeeding;
7. Patients voluntarily joined the study and signed informed consent;

Exclusion Criteria:

1. Patients have evidence of metastatic breast cancer, or inflammatory breast cancer;
2. Patients previously received antineoplastic therapy or radiotherapy for any malignancy, excluding cured malignancies such as cervical carcinoma in situ, basal cell carcinoma, or squamous carcinoma;
3. Patients received any other anti-tumor therapy at the same time, including endocrine therapy, bisphosphonates or immunotherapy;
4. Patients have major surgical procedures unrelated to breast cancer within 4 weeks before the first medication, or not fully recovered from surgical procedures;
5. Clinically significant pulmonary or cardiovascular disease;
6. Failure to swallow, chronic diarrhea, intestinal obstruction, or presence of other factors affecting drug administration and absorption;
7. Known to be allergic to any study drug or any of its excipients;
8. History of immunodeficiency, including HIV-positive, or other acquired or congenital immunodeficiency diseases, or history of organ transplantation;
9. Pregnant and lactating women;
10. Patients with serious concomitant diseases or other comorbidities that will interfere with the planned treatment, or any other condition that is not suitable for participation assessed by investigator.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-07-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) Tumours (RECIST) v1.1 | During 24 weeks of the neoadjuvant treatment
  Objective Response Rate (ORR) according to Response Evaluation Criteria in Solid

SECONDARY OUTCOMES:
Incidence of Adverse Events | from consent to 28 days after last dose
  Evaluate the nature, incidence and severity of SHR-A1811 adverse events according to CTCAE 5.0
Residual cancer burden (RCB) | At the time of surgery
  Residual cancer burden (RCB)
Pathological complete response | At the time of surgery
  pCR: ypT0/is ypN0
Event-free survival (EFS) | 5 years
  EFS was defined as the time from randomization to any of the following events: disease progression during neoadjuvant therapy, local or distant recurrence, second primary malignancy (breast or other cancer), or death from any cause
Disease-free survival (DFS) | 5 years
  Disease-free Survival, From the date of surgery to the first local, regional, contralateral or distant recurrence, and death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Zhenzhen Liu, PhD, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No